CLINICAL TRIAL: NCT04895163
Title: Acute Appendicitis in Foreign Workers of Northern Israel: a Retrospective Cohort Study
Brief Title: Acute Appendicitis in Foreign Workers of Northern Israel
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Uri Kaplan , MD, Acting head of bariatri center, Head of GEJ surgical unit, HaEmek Medical Center, Israel
Other Study IDs: 106-18-EMC
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Surgery
Keywords: Acute appendicitis; Foreign workers; Complicated appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Foreign workers: Foreign workers aged 18-50 who were admitted to our institution between January 1st, 2013 and October 31st, 2018, with the diagnosis of acute appendicitis.
  Interventions: Procedure: Laparoscopic appendectomy
- Local patients: Local patients aged 18-50 who were admitted to our institution between January 1st, 2013 and October 31st, 2018, with the diagnosis of acute appendicitis.
  Interventions: Procedure: Laparoscopic appendectomy

INTERVENTIONS:
Procedure: Laparoscopic appendectomy — Laparoscopic appendectomy performed for acute appendicitis

SUMMARY:
To Compare the outcome to acute appendicitis in foreign workers to the native patients.

DETAILED DESCRIPTION:
This is a retrospective case-control study. The investigators identified all patients aged 18-50 who were admitted to our institution between January 1st, 2013 and October 31st, 2018, with the diagnosis of acute appendicitis. The study group included all foreign workers and the control group was age, sex, and co-morbidities matched group from the local population. The investigators compared time to presentation, admission parameters and disease outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-50 who were admitted to our institution between January 1st, 2013 and October 31st, 2018, with the diagnosis of acute appendicitis

Exclusion Criteria:

* Pregnant women
* Patient whose pathology report of the appendix was normal

Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 18-50 who were admitted to our institution between January 1st, 2013 and October 31st, 2018, with the diagnosis of acute appendicitis
Sampling Method: Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Percent of complicated disease | 1 month
  amount of cases defined as complicated acute appendicitis

CONTACTS AND LOCATIONS:
Locations (1):
- Emek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: Undecided